CLINICAL TRIAL: NCT04697056
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ANB019 in the Treatment of Subjects With Ichthyosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Participants With Ichthyosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative Reason
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-206; 2020-003476-41 (EudraCT Number)
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-11

CONDITIONS: Ichthyosis
Keywords: IL-36 Receptor; Interleukin 36; Imsidolimab
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imsidolimab (Experimental): Participants received a starting dose of 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
  Interventions: Drug: Imsidolimab
- Placebo (Placebo Comparator): Participants received imsidolimab matching placebo on Day 1 and thereafter, every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
  Interventions: Biological: placebo

INTERVENTIONS:
Drug: Imsidolimab — Humanized Monoclonal Antibody
  Other Names: ANB019
  Arms: Imsidolimab
Biological: placebo — placebo
  Arms: Placebo

SUMMARY:
Efficacy and Safety of imsidolimab in Participants with Ichthyosis

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of imsidolimab compared with placebo in adolescent and adult participants with ichthyosis. This study will also characterize the pharmacokinetic (PK) profile of imsidolimab and explore the immune response to imsidolimab in participants with ichthyosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ichthyosis
* IASI total score ≥ 18, erythema score ≥ 2
* Participant has been using emollient daily for at least 1 week prior to Day 1 and agrees to continue using that same emollient daily at the same frequency throughout the study

Exclusion Criteria:

* A participant with ichthyosis vulgaris, X-linked ichthyosis, or lamellar ichthyosis will be excluded.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Site 106, Palo Alto, California
  - Site 104, New Haven, Connecticut
  - Site 112, Miami, Florida
  - Site 101, Chicago, Illinois
  - Site 102, Columbus, Ohio
  - Site 107, San Antonio, Texas
  - Site 105, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with confirmed diagnosis of ichthyosis by genetic testing of ichthyosis were enrolled into the study.
Pre-assignment Details: 7 participants were screened for eligibility and 5 participants were randomized into the study.
Groups:
- Placebo: Participants received imsidolimab matching placebo on Day 1 and thereafter every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
Period: Overall Study
Arm/Group | Imsidolimab | Placebo
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Termination of the participant participation by the Investigator or Sponsor | 4 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set included all randomized participants.
Groups:
- Imsidolimab: Participants received a starting dose of 400 mg of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Imsidolimab | Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (20.15) | 66.0 | 44.4 (21.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ichthyosis Area Severity Index (IASI) Total Score at Week 16
Description: IASI quantified the severity of participants ichthyosis based on severity of erythema/scaling & percentage of body surface area (BSA) affected. Degree of erythema & scaling scored from 0 (none) to 4 (very severe) for each of 4 body regions (BR) [A1: head & neck (H&N), A2: upper limbs (UL), A3: trunk (T), A4: lower limbs (LL)]. Percentage of BSA involved for each BR (B1: % in H&N, B2: % in UL, B3: % in T, B4: % in LL). Percentage involvement was assigned numerical value(0= 0, 1%-9%= 1, 10%-29%= 2, 30%-49%= 3, 50%-69%= 4, 70%-89%= 5, 90%-100%= 6).Total extent was determined using multiplier considering % of total BSA by each BR (C1= 0.1 for H&N; C2= 0.2 for UL; C3= 0.3 for T; C4= 0.4 for LL).
  IASI-Erythema (E)= A1E x B1 x C1 + A2E x B2 x C2 + A3E x B3 x C3 + A4E x B4 x C4 (score 0 to 24) IASI-Scaling (S)= A1S x B1 X C1 + A2S x B2 x C2 + A3S x B3 x C3 + A4S x B4 x C4 (score 0 to 24) IASI total score= IASI-E + IASI-S score ranged from 0 - 48, higher score indicated worse disease state.
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in IASI Total Score at Week 16
Description: IASI quantified the severity of participants ichthyosis based on severity of erythema/scaling, & percentage of BSA affected. Degree of erythema & scaling scored from 0 (none) to 4 (very severe) for each of 4 BR (A1: H&N, A2: UL, A3: T, A4: LL). Percentage of BSA involved for each BR (B1: % in H&N, B2: % in UL, B3: % in T, B4: % in LL). Percentage involvement was assigned numerical value (0= 0, 1%-9%= 1, 10%-29%= 2, 30%-49%= 3, 50%-69%= 4, 70%-89%= 5, 90%-100%= 6). Total extent was determined using a multiplier considering % of total BSA by each BR (C1= 0.1 for H&N; C2= 0.2 for UL; C3= 0.3 for T; C4= 0.4 for LL).
  IASI-E= A1E x B1 x C1 + A2E x B2 x C2 + A3E x B3 x C3 + A4E x B4 x C4 (score 0 to 24)
  IASI-S= A1S x B1 X C1 + A2S x B2 x C2 + A3S x B3 x C3 + A4S x B4 x C4 (score 0 to 24)
  IASI total score= IASI-E + IASI-S score ranged from 0 - 48, higher score indicated worse disease state.
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving an Improvement of 50% From Baseline in IASI (IASI50) at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in IASI-E Scores at Week 16
Description: IASI quantified the severity of participants ichthyosis based on severity of erythema/scaling, & percentage of BSA affected. Degree of erythema & scaling scored from 0 (none) to 4 (very severe) for each of 4 BR (A1: H&N, A2: UL, A3: T, A4: LL). Percentage of BSA involved for each BR (B1: % in H&N, B2: % in UL, B3: % in T, B4: % in LL). Percentage involvement was assigned numerical value (0= 0, 1%-9%= 1, 10%-29%= 2, 30%-49%= 3, 50%-69%= 4, 70%-89%= 5, 90%-100%= 6). Total extent was determined using a multiplier considering % of total BSA by each BR (C1= 0.1 for H&N; C2= 0.2 for UL; C3= 0.3 for T; C4= 0.4 for LL).
  IASI-E= A1E x B1 x C1 + A2E x B2 x C2 + A3E x B3 x C3 + A4E x B4 x C4
  IASI-E score ranged from 0 - 24, higher score indicated worse disease state.
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in IASI-S Scores at Week 16
Description: IASI quantified the severity of participants ichthyosis based on severity of erythema/scaling, & percentage of BSA affected. Degree of erythema & scaling scored from 0 (none) to 4 (very severe) for each of 4 BR (A1: H&N, A2: UL, A3: T, A4: LL). Percentage of BSA involved for each BR (B1: % in H&N, B2: % in UL, B3: % in T, B4: % in LL). Percentage involvement was assigned numerical value (0= 0, 1%-9%= 1, 10%-29%= 2, 30%-49%= 3, 50%-69%= 4, 70%-89%= 5, 90%-100%= 6). Total extent was determined using a multiplier considering % of total BSA by each BR (C1= 0.1 for H&N; C2= 0.2 for UL; C3= 0.3 for T; C4= 0.4 for LL).
  IASI-S= A1S x B1 X C1 + A2S x B2 x C2 + A3S x B3 x C3 + A4S x B4 x C4
  IASI-S score ranged from 0 - 24, higher score indicated worse disease state.
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in IASI-E Scores at Week 16
Description: as for outcome 4
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Groups:
- Placebo: Participants received imsidolimab matching placebo on day 1 and thereafter every four weeks (days 29, 57 and 85) by subcutaneous injection.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in IASI-S Scores at Week 16
Description: as for outcome 5
Time Frame: Baseline and Week 16
Population: Due to early study termination before the primary time point, efficacy data was not collected, therefore, not analyzed.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of study treatment that did not necessarily have a causal relationship with this treatment. An AE was considered "serious" if there was any of the following outcomes: death, life-threatening adverse event, Inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, other important medical events. An adverse event was considered TE if the date of onset was during or after first dose of study treatment, or if the AE present at baseline worsened in either intensity or frequency after first dose of study treatment.
Time Frame: From first dose up to study termination (maximum up to 9.4 weeks)
Population: Safety analysis set included all randomized participants who received at least 1 dose of imsidolimab or placebo.
Measure: Number; unit: participants
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 4 | 1
participants
  Any TEAEs | 1 | 1
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to study termination (maximum up to 9.4 weeks)
Description: Safety analysis set included all randomized participants who received at least 1 dose of imsidolimab or placebo.
Groups:
- Imsidolimab: Participants received a starting dose of 400 mg of imsidolimab on Day 1 followed by 200 mg imsidolimab every four 4 (Days 29, 57 and 85) by subcutaneous injection.
- Placebo: Participants received imsidolimab matching placebo on Day 1 and thereafter every four 4 (Days 29, 57 and 85) by subcutaneous injection.
Arm/Group | Imsidolimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 1/4 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imsidolimab (N=4) | Placebo (N=1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
As a result of insufficient recruitment of participants, this study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT04697056/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04697056/SAP_001.pdf